CLINICAL TRIAL: NCT00639769
Title: Phase II Trial of Irinotecan Plus Cisplatin in Patients With Recurrent or Metastatic Squamous Carcinoma of the Head and Neck
Brief Title: Irinotecan and Cisplatin in Treating Patients With Recurrent or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Murphy, MD, Professor of Medicine; Director, Cancer Supportive Care Program; Director, Head and Neck Research Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC HN 0164; VU-VICC-HN-0164; VU-VICC-01-0847
Record Dates: First submitted 2008-03-19; First posted 2008-03-20 (Estimated); Results first posted 2011-12-07 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; untreated metastatic squamous neck cancer with occult primary; recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; salivary gland squamous cell carcinoma; stage IV salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Cisplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic Intervention (Experimental)
  Interventions: Drug: cisplatin; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: cisplatin — Starting dose 30 mg/m2 Dose level -1 20 mg/m2
  Other Names: Platinol,Platinol-AQ,cisdamminedichloroplatinum(II),kCDDP,DDP,DACP,cisplatinum,platinum
Drug: irinotecan hydrochloride — 50 mg/m2 IV over 60 minutes, plus Cisplatin 30mig/m2 IV, repeated weekly for two weeks. followed by a one-week rest. This 3-week schedule given two times to equal one 6-week cycle. Maximum of 6 cycles.
  Other Names: CPT-11

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: To determine if CPT-11 given together with cisplatin is effective in treating recurrent or metastatic head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the efficacy of irinotecan hydrochloride and cisplatin in patients with local-regionally recurrent or metastatic squamous cell carcinoma of the head and neck.
* Evaluate the toxicity of irinotecan hydrochloride and cisplatin in these patients.
* Determine the palliative effect of irinotecan hydrochloride and cisplatin on head and neck cancer symptoms using the Vanderbilt Cancer Center (VICC) Head and Neck Cancer Symptom Survey.

OUTLINE: Patients receive irinotecan hydrochloride IV over 60 minutes and cisplatin IV on days 1, 8, 22, and 29. Treatment repeats every 6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients complete the Vanderbilt Cancer Center (VICC) Head and Neck Cancer Symptom Survey at baseline, before each course, at the completion of study therapy, and then at each follow-up visit.

After completion of study therapy, patients are followed every 6 weeks for 1 year and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the head and neck that is considered incurable with surgery or radiotherapy
* Meets one of the following criteria:

  * Previously untreated disease

    * Newly diagnosed disease with distant metastases
  * Recurrent or persistent disease

    * Local-regional recurrence/persistence or distant metastases after initial treatment with surgery or radiotherapy

      * No locally advanced unresectable disease that was not previously treated with radiotherapy
* Bidimensionally measurable disease

  * If the only measurable disease is within the radiotherapy port, there must be biopsy-proven recurrence ≥ 8 weeks after the completion of radiotherapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Creatinine clearance ≥ 50 mL/min
* SGOT ≤ 3 times upper limit of normal
* Serum bilirubin < 1.5 mg/dL
* Granulocytes ≥ 1,500/mm ^3
* Platelet count > 100,000/mm^3
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant detectable infection
* No co-morbid disease unless under adequate control
* No other cancer within the past 3 years except basal cell or squamous cell skin cancer or early-stage prostate cancer

Exclusion Criteria:

-Pregnant or lactating women

Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from any prior major surgery
* No prior chemotherapy for recurrent or metastatic disease

  * Patients who completed neoadjuvant, concurrent, or adjuvant chemotherapy ≥ 3 months prior to recurrence will be considered chemotherapy-naive
  * Patients who completed neoadjuvant, concurrent, or adjuvant chemotherapy < 3 months prior to recurrence will be considered chemotherapy failures
* No prior therapy with topotecan or irinotecan hydrochloride
* At least 4 weeks since prior biologic therapy (e.g., interleukin-2, interferon, megestrol acetate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2002-02; Primary Completion 2007-05 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A. Murphy, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (8):
- United States (8):
  - Central Georgia Hematology Oncology Associates, P.C., Macon, Georgia
  - Erlanger Health System, Chattanooga, Tennessee
  - Jackson-Madison County Hospital, Jackson, Tennessee
  - East Tennessee State University, Johnson City, Tennessee
  - Center for Biomedical Research, Knoxville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - VA Tennessee Valley Healthcare Center, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Result] Gilbert J, Cmelak A, Shyr Y, Netterville J, Burkey BB, Sinard RJ, Yarbrough WG, Chung CH, Aulino JM, Murphy BA. Phase II trial of irinotecan plus cisplatin in patients with recurrent or metastatic squamous carcinoma of the head and neck. Cancer. 2008 Jul 1;113(1):186-92. doi: 10.1002/cncr.23545. PMID 18484593

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period = 2/27/2002 through 5/9/2006
Pre-assignment Details: A total of 41 people signed consent to take part in this study, of those, 1 was determined to be ineligible.
Groups:
- Therapeutic Intervention: Cisplatin, Starting dose 30 mg/m2 Dose level -1 20 mg/m2; Irinotecan, Starting Dose 50 mg/m2, Dose level -1 40 mg/m2
Period: Overall Study
Arm/Group | Therapeutic Intervention
Started | 40
Completed | 0
Not Completed | 40
Not completed — Death | 2
Not completed — Adverse Event | 7
Not completed — Lack of Efficacy | 1
Not completed — Disease progression | 26
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 58 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Patient Response
Description: Number of patients in each response category according to RECIST criteria: Progressive disease (PD): >=20% increase in sum of longest diameter (LD) of target lesion(s), taking as reference smallest sum LD recorded since treatment started. Complete response (CR): disappearance of all target lesions. Partial response (PR): >=30% decrease in sum of LD of target lesion(s), taking as reference baseline sum LD. Stable disease (SD): neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD.
Time Frame: 6 weeks after last chemotherapy treatment
Population: Analysis was per protocol (7 patients did not receive a full cycle of treatment, and 1 patient was censored for incomplete records)
Measure: Number; unit: participants
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 32
participants
  Partial Response | 11
  Progressive Disease | 15
  Stable Disease | 6
  Complete response | 0

2. Secondary Outcome: Number of Patients With Each Worst-grade Toxicity
Description: Number of patients with worst-grade toxicity response of each grade (grade 1 to 5) following NCI Common Toxicity Criteria, with grade 1=mild adverse event; 2=moderate adverse event; 3=severe and undesirable adverse event; 4=life-threatening or disabling adverse event; 5=death
Time Frame: 6 weeks after last chemotherapy
Measure: Number; unit: participants
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 40
participants
  No. of patients with worst-grade toxicity of 1 | 2
  No. of patients with worst-grade toxicity of 2 | 12
  No. of patients with worst-grade toxicity of 3 | 21
  No. of patients with worst-grade toxicity of 4 | 10
  No. of patients with worst-grade toxicity of 5 | 1

ADVERSE EVENTS:
Arm/Group | Therapeutic Intervention
Serious Adverse Events (participants affected / at risk) | 27/40
Other Adverse Events (participants affected / at risk) | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic Intervention (N=40)
Abdominal distention (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 13 (13)
Depressed level of consciouness (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 11 (11)
Dysphagia - esophageal (related to radiation) (Gastrointestinal disorders) | 1 (1)
Dysphagia, esophagitis, odynophagai (Gastrointestinal disorders) | 3 (3)
Facial cellulitis (Infections and infestations) | 2 (2)
Fatigue (General disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Hemoglobin decreased (Investigations) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Illeus (Gastrointestinal disorders) | 1 (1)
Infected gastrocutaneous fistula (Gastrointestinal disorders) | 1 (1)
Leukocytes (WBC 1.3) (Investigations) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (10)
Neutrophil count decreased (Investigations) | 6 (6)
Platelet count decreased (Investigations) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Post-nasal drip (General disorders) | 1 (1)
Right shoulder pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Subacute fx of L1 vertebral body (Musculoskeletal and connective tissue disorders) | 1 (1)
Thromboembolism (Vascular disorders) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 13 (13)
Weakness (General disorders) | 2 (2)
White blood cell decrease (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes